CLINICAL TRIAL: NCT01963273
Title: Video Assisted Ablation of Pilonidal Sinus. Evaluation of Safety and Efficacy of a New Minimally Invasive Technique
Brief Title: Video Assisted Ablation of Pilonidal Sinus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Francesco Milone, Professor, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5082; Surgery
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

ARMS (1):
- pilonidal sinuses (Experimental): All consecutive patients with diagnosis of chronic sacrococcygeal pilonidal sinus will be screened for the enrollment in our study.
  Interventions: Procedure: Video Assisted Ablation of Pilonidal Sinus

INTERVENTIONS:
Procedure: Video Assisted Ablation of Pilonidal Sinus

SUMMARY:
The investigators supposed that the complete video assisted ablation of pilonidal sinus (VAAPS) could be an effective minimally invasive treatment of pilonidal sinus. This new minimally invasive treatment allows the identification of the sinus cavity with its lateral tracks, the destruction and the removal of all infected tissue and the removing of any hair.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of chronic pilonidal sinus

Exclusion Criteria:

Inability to consent to the study Recurrent pilonidal sinus after an outmidline technique

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Infection | 1 month
  Wound infection was defined as redness and/or oedema of the skin and/or discharge

SECONDARY OUTCOMES:
Recurrence | 1 year
  Recurrence can be divided into two groups: early and late. Early recurrence is usually due to failure to identify one or more sinuses. Late recurrence is usually due to secondary infection caused by residual hair or debris that was not removed at operation, inadequate wound care or insufficient attention to depilation

OTHER OUTCOMES:
time off work | 1 month
Time to sitting on toilet without pain | 1 month
satisfaction | 6 months
  Satisfaction Scores on the Visual Analog Scale
Aesthetic appearance | 6 months
  Aesthetic appearance on a 3 points scale of good fair and bad
Pain | 1 day, 1 week and 1 month
  Pain Scores on the Visual Analog Scale
time to walk without pain | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Milone Francesco, Naples, Italiy, Italy

REFERENCES:
- [Derived] Milone M, Fernandez LM, Musella M, Milone F. Safety and Efficacy of Minimally Invasive Video-Assisted Ablation of Pilonidal Sinus: A Randomized Clinical Trial. JAMA Surg. 2016 Jun 1;151(6):547-53. doi: 10.1001/jamasurg.2015.5233. PMID 26819186